CLINICAL TRIAL: NCT00833352
Title: Comparison of Right Ventricular Septal and Right Ventricular Apical Pacing in Patients Receiving a CRT-D Device
Acronym: SEPTAL-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guidant Corporation (Industry)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEPTAL CRT 0408
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Systolic Heart Failure; Ventricular Tachycardia; Ventricular Fibrillation
MeSH Terms: conditions — Heart Failure, Systolic; Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Right ventricular lead located in Mid Septum
  Interventions: Device: CRT-D Therapy
- 2 (Active Comparator): Right ventricular lead located in Apex
  Interventions: Device: CRT-D Therapy

INTERVENTIONS:
Device: CRT-D Therapy — Implant of a defibrillator with cardiac resynchronization therapy to detect and terminate ventricular arrhythmias and resynchronize ventricles.
  Other Names: Endotak Reliance G and SG

SUMMARY:
This prospective, randomized, single blind, multi-centre study will examine the effect of the right ventricular (RV) lead location in patients implanted with a cardiac resynchronization defibrillator.

1. Purpose :

   To compare the effect of RV mid-septal (RVS) versus RV apical (RVA) lead location on left ventricular reverse remodeling in patients indicated for cardiac resynchronization therapy device (CRT-D) over a period of 6 months and to evaluate the clinical outcome of the RVS versus RVA pacing, over a period of 12 months.
2. Objectives:

The primary objective is to demonstrate that there is no difference between the two groups (RVA vs. RVS) in the change of left ventricular end systolic volume (LVESV), between baseline and 6 months.

The secondary objectives are to evaluate the percentage of "echo-responders" plus additional clinical and safety outcomes.

This prospective, randomized, multi-centre, single-blind with 2 parallel arms, non-inferiority study will be conducted in approximately 25 study centres in Europe. The patients will be randomized in a 1:1 ratio. A maximum of 416 patients will be enrolled in this study.

All eligible patients will be followed through baseline, randomisation, pre discharge, 1, 6 and 12 months post-implant. Enrolment is expected to be completed in 18 months. The total duration of the study is expected to be approximately 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Accepted CRT indication according to ESC with

  1. Documented LVEF </= 35% in last 3 months
  2. Documented LVEDD ≥ 55 mm or LVEDD > 30 mm/m2, or LVEDD >30 mm/m (height) in last 3 months
  3. QRS ≥120 ms documented on ECG recording during hospitalisation
  4. NYHA Class III or ambulatory class IV stable for the last month previous enrolment
* Or the previous criteria 1 and 2 and a transient episode in NYHA class III or IV with prior HF hospitalization or intravenous decongestive therapy (IV diuretics, IV neseritide or IV inotropes) in an "out-patient" setting within the year previous enrolment and stabilization to NYHA class II for the last month with a QRS ≥150 ms documented on ECG recording during hospitalisation
* ICD indication (class I or II A)
* Optimal and stable medication for at least one month (except for diuretics stable for minimum 1 week) based on ESC guidelines before the enrolment
* Chronic heart failure (> 3 months) stable for the last month previous enrolment
* Stable sinus rhythm at the enrolment
* Willing and capable of providing informed consent

Exclusion Criteria

* Defibrillation testing not planned during the implant procedure due to a poor haemodynamic or clinical status or other reasons
* Have persistent atrial fibrillation (AF) or atrial flutter (i.e, can be terminated with medical intervention, but does not terminate spontaneously) within 1 month prior inclusion
* Documented AF within 1 month prior enrolment
* Life expectancy < 12 months or expected to undergo heart transplant within the next 12 months
* Uncontrolled blood pressure (Systolic BP > 160 mmHg or Diastolic BP > 85 mmHg)
* Hospitalization for HF or intravenous inotropic drug treatment within 1 month prior enrolment
* Cardiac surgery, per cutaneous transluminal angioplasty (PTCA), myocardial infarction (MI), unstable or severe angina or stroke during last 3 months prior enrolment
* Previously implanted pacemaker or ICD
* Uncorrected primary valvular disease
* Prosthetic tricuspid valve
* Nursing women or of childbearing potential who are, or might be pregnant at the time of the study
* Enrolled in any on-going study (including pharmacologic trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
left ventricular end systolic volume (LVESV) | 6 months

SECONDARY OUTCOMES:
left ventricular end systolic volume | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Leclercq, MD, Principal Investigator — Hopital Pontchaillou - Rennes- France; Ignacio Fernández Lozano, MD, Principal Investigator — Hospital Puerta de Hierro - Madrid - Spain
Locations (26):
- France (17):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hôpital Louis Pradel, Bron
  - Centre Hospitalier Universitaire de Grenoble- Hôpital Albert Michalon, Grenoble
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Hôpital Saint Joseph, Marseille
  - Centre Hospitalier Universitaire de Marseille- Hôpital La Timone, Marseille
  - Centre Hospitalier Universitaire de Montpellier- Hôpital Arnaud de Villeneuve, Montpellier
  - Nouvelles Cliniques Nantaises, Nantes
  - Centre Hospitalier Régional d'Orléans- Hôpital La Source, Orléans
  - Hôpital La Pitié Salpétrière, Paris
  - Centre Hospitalier Universitaire Haut Levêque, Pessac
  - Centre Hospitaler Universitaire Pontchaillou, Rennes
  - Centre Hospitalier Universitaire-Charles Nicolle, Rouen
  - Centre Cardiologique du Nord, Saint-Denis
  - Centre Hospitalier Universitaire - Hôpital Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
  - Centre Hospitalier Universitaire de Nancy- Hôpital Brabois, Vandœuvre-lès-Nancy
- Spain (9):
  - Hospital general de Alicante, Alicante
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Puerta de Hierro, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Virgen de la salud de Toledo, Toledo
  - Hospital La Fe, Valencia
  - Hospital Universitario Río Hortega, Valladolid

REFERENCES:
- [Derived] Leclercq C, Sadoul N, Mont L, Defaye P, Osca J, Mouton E, Isnard R, Habib G, Zamorano J, Derumeaux G, Fernandez-Lozano I; SEPTAL CRT Study Investigators. Comparison of right ventricular septal pacing and right ventricular apical pacing in patients receiving cardiac resynchronization therapy defibrillators: the SEPTAL CRT Study. Eur Heart J. 2016 Feb 1;37(5):473-83. doi: 10.1093/eurheartj/ehv422. Epub 2015 Sep 15. PMID 26374852